CLINICAL TRIAL: NCT05902585
Title: Usefulness of Virtual Reality in the Management of Pain Associated With Venipuncture in Pediatrics: a Multi-center Randomized Clinical Trial
Brief Title: Virtual Reality in the Management of Pain in Pediatrics: a Multi-center Randomized Clinical Trial (RealPED)
Acronym: RealPED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Principal Investigator, Raquel Gil Piquer, Principal investigator, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 37/2021
Record Dates: First submitted 2023-05-15; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Virtual Reality; Pediatric ALL; Pain, Procedural
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Pain, Procedural

STUDY DESIGN:
Intervention Model Description: Patients are randomized in a 1:1 ratio to the intervention group (use of virtual reality during blood collection) and the control group (usual care). The randomization sequence is different for each participating center.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): In this arm, the analysis will be done in the usual way (for example, distracting with questions).
- Virtual reality (Active Comparator): In this arm, the analysis will be done while the children use virtual reality.
  Interventions: Behavioral: Virtual reality

INTERVENTIONS:
Behavioral: Virtual reality — In the virtual reality group, patients will view a video with the virtual reality glasses from the beginning to the end of the venipuncture.
  Arms: Virtual reality

SUMMARY:
The goal of this clinical trial is to test if the use of virtual reality glasses reduces the pain and anxiety that children feel when they perform a blood test.

Children between 7 and 12 years old from 5 health centers and 2 hospitals will participate, and the children will be divided into two groups. In the control group, the analysis will be done in the usual way (for example, distracting with questions) and in the intervention group, the analysis will be done while the children use virtual reality.

The satisfaction of parents and nursing will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Children between 7 and 12 years old who attend participating centers for scheduled blood tests.
* Consent to participate by signing the informed consent.

Exclusion Criteria:

* Children younger than 7 years old.
* Children older than 12 years old.
* Children that don't sign the informed consent.
* Children with psychomotor and neurocognitive delay.
* Children with visual or hearing impairment.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 83 (Actual)
Dates: Start 2022-02-26 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
Pain associated with venipuncture | 1 day: The day of the venipuncture
  Visual analog scale: From 1 to 10. 1 implies minimal pain and 10 unbearable pain.
Anxiety | 1 day: The day of the venipuncture
  Groningen distress scale: From 1 to 5. 1 implies a non-anxious patient and 5 a very anxious patient.

SECONDARY OUTCOMES:
Number of attempts for analytics | 1 day: The day of the venipuncture
  1, 2, 3, 4, or 5
Time required for analysis | 1 day: The day of the venipuncture
  Minutes
Difficulty level of the technique | 1 day: The day of the venipuncture
  Easy, normal or difficult
Parents satisfaction | 1 day: The day of the venipuncture
  1 = unsatisfied 10 = very satisfied
Nurse anxiety | 1 day: The day of the venipuncture
  1 = totally calm 10 = very anxious

OTHER OUTCOMES:
Pacient age at the moment of venipuncture | Before venipuncture
  In years
Pacient sex | Before venipuncture
  Male or female
Venipuncture in the last 6 months | Before venipuncture
  Venipuncture in the last 6 months
Parental presence at the moment of venipuncture | 1 day: The day of the venipuncture
  Yes or not

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Gil Piquer, Principal Investigator — Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Locations (6):
- Spain (6):
  - Centre de Salut de Castelló, Castellon, Valencia
  - Centre de Salut de Carcer, Càrcer, Valencia
  - Centre de Salut de Pobla Llarga, La Pobla Llarga, Valencia
  - Hospital General de Onteniente, Ontinyent, Valencia
  - Centre de Salut de Xàtiva, Xàtiva, Valencia
  - Hospital Lluís Alcanyís, Xàtiva, Valencia

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-22): https://cdn.clinicaltrials.gov/large-docs/85/NCT05902585/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-22): https://cdn.clinicaltrials.gov/large-docs/85/NCT05902585/ICF_001.pdf